CLINICAL TRIAL: NCT04664179
Title: Constitutive IL7 (C7R) Modified EBV Specific T-Lymphocytes for Treatment of EBV-Positive Lymphoma
Brief Title: EBV Specific T-Lymphocytes for Treatment of EBV-Positive Lymphoma
Acronym: CILESTE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bilal Omer, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-47906 CILESTE; P50CA126752 (NIH)
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: EBV-Related Hodgkin Lymphoma; EBV-Related Lymphoproliferative Disorder; EBV Related Non-Hodgkin's Lymphoma
Keywords: non-Hodgkin's Lymphoma; EBV (associated)-T/NK-lymphoproliferative disease; EBV SPECIFIC T-LYMPHOCYTES; EBV; Hodgkin's Lymphoma; lymphoma relapse
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Epstein-Barr Virus Infections; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Treatment without lymphodepletion chemotherapy (Experimental): C7R-EBVSTs
  Group B will be activated if only limited expansion and clinical efficacy is observed in Group A
  Interventions: Biological: Dose Level 1A: 2 x 10^7 cells/m2; Biological: Dose Level 2A: 6 x 10^7 cells/m2; Biological: Dose Level 3A: 2 x 10^8 cells/m2
- Arm B: Treatment with lymphodepletion chemotherapy (Experimental): C7R-EBVSTs with lymphodepletion chemotherapy
  Interventions: Biological: Dose Level 2B: 6 x 10^7 cells/m2; Biological: Dose Level 3B: 2 x 10^8 cells/m2

INTERVENTIONS:
Biological: Dose Level 1A: 2 x 10^7 cells/m2 — 2 x 10^7 cells/m2
  Arms: Arm A: Treatment without lymphodepletion chemotherapy
Biological: Dose Level 2A: 6 x 10^7 cells/m2 — 6 x 10^7 cells/m2
  Arms: Arm A: Treatment without lymphodepletion chemotherapy
Biological: Dose Level 2B: 6 x 10^7 cells/m2 — 6 x 10^7 cells/m2
  Arms: Arm B: Treatment with lymphodepletion chemotherapy
Biological: Dose Level 3B: 2 x 10^8 cells/m2 — 2 x 10^8 cells/m2
  Arms: Arm B: Treatment with lymphodepletion chemotherapy
Biological: Dose Level 3A: 2 x 10^8 cells/m2 — 2 x 10^8 cells/m2
  Arms: Arm A: Treatment without lymphodepletion chemotherapy

SUMMARY:
This study is for patients that have a type of lymph gland disease called Hodgkin or non-Hodgkin Lymphoma or T/NK-lymphoproliferative disease which has come back or has not gone away after treatment, including the best treatment the investigators know for these diseases.

Some patients with Lymphoma or T/NK-lymphoproliferative disease show signs of virus that is sometimes called Epstein Barr virus (EBV) that causes mononucleosis or glandular fever ("mono") before or at the time of their diagnosis. EBV is found in the cancer cells of up to half the patients with Hodgkin's and non-Hodgkin Lymphoma, suggesting that plays a role in causing Lymphoma. The cancer cells (in lymphoma) and some immune system cells infected by EBV are able to hide from the body's immune system and escape destruction.

T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. T cells have been used to treat patients with cancers. T cells, that have been trained to kill EBV infected cells can survive in the blood and affect the tumor. The investigators have treated over 80 people on studies using T cells to target these diseases. About half of those patients who had disease at the time they got the cells had responses including some patients with complete responses.

The investigators think that if T cells are able to last longer in the body, they may have a better chance of killing EBV and EBV infected tumor cells. Therefore, in this study the investigators will add a new gene to the EBV T cells that can cause the cells to live longer called C7R. The investigators know that T cells need substances called cytokines to survive and the cells may not get enough cytokines after infusion into the body. The investigators have added the gene C7R that gives the cells a constant supply of cytokine and helps them to survive for a longer period of time.

The purpose of this study is to find the largest safe dose of C7R-EBV T cells, and additionally to evaluate how long they can be detected in the blood and what affect they have on cancer.

DETAILED DESCRIPTION:
The patient will donate blood in order to make C7R-EBV T cells. Depending on how long ago the cells were generated, they have been frozen. To get the C7R to be made by the T-cell, the investigators inserted a gene into the T-cell. This is done using certain parts of a virus (known as a retrovirus) that can carry the gene into the T cells. Because patients receive cells with a new gene in them, they will befollowed for a total of 15 years to see if there are any long term side effects of gene transfer.

When they are enrolled in this study, patients are assigned a dose of C7R EBV T cells. The assigned dose of cells is based on body weight and height. Patients will receive the C7R EBV T cells and may also receive cyclophosphamide and fludarabine (these are standard chemotherapy medicines). The chemotherapy medicines may be given before the T cells to make space in the blood for the T cells to grow after receiving them.

If a patient receives chemotherapy medicines, these drugs will be given through an i.v. needle inserted in the patient's vein or central line) for 2 days and then fludarabine alone on the third day. The patient will be given an injection of C7R EBV T cells into the vein through an IV line at the assigned dose.

Patients may receive Benadryl and Tylenol. The infusion will take between 1 and 10 minutes. The investigators will then monitor the patient in the clinic or hospital for about 2 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. Patients should plan to stay in Houston for up to 2 weeks after the infusion so the investigators can monitor them for side effects.

Patients will have follow-up visits with the clinic (at scheduled visits weeks 2 and 6, and nursing follow-up at weeks 1, 2, 4, and 6; months 3, 6, 9, and 12; and annually for the next 15 years). Patients will have scheduled disease evaluations after the T-cell injection (at week 6 +/- 2 weeks and then as clinically needed). After the disease re-evaluation, if the patient's disease has not gotten worse, or if in the future it seems he/she might benefit, they may be eligible to receive one additional dose of the T cells. The dose will be at the same dose level as the patient's first infusion and separated by at least 6 weeks such that the investigators can make sure that the patient has no severe side effects between infusions. If the patient receives an additional dose of C7R EBV T-cells, they will need to stay in Houston for up to 2 weeks after the infusion as well so the investigators can monitor them for side effects.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies. The investigators will use the imaging studies that have been used in the past to best assess the patient's tumor (Computer Tomogram (CT) or Magnetic Resonance Imaging (MRI), and Positron Emission Tomography (PET/CT) and/or Bone Scan).

Medical tests during and after treatment--

The patient will receive standard medical tests when they are getting the infusions and afterwards:

* Physical exams
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies approximately 6 weeks after the infusion.

To learn more about the way the C7R EBV T cells are working and how long they last in the body, an extra amount of blood will be obtained on the day that chemotherapy starts, the day of the T-cell infusion(s) and at the end of the T-cell infusion(s), 1, 2, 4, 6 weeks after the T-cell infusion(s) and every 3 months for the 1st year, and annually for the next 15 years and possibly at additional time points. The amount of blood taken will be based on the patient's weight with up to a maximum of 60 mL (12 teaspoons) of blood to be obtained at any one time. For children, the total amount of blood drawn will not be more than 3 mL (less than 1 teaspoon) per 1 kg (2 lbs) of body weight on any one day. This volume is considered safe, but may be decreased if the patient is anemic (have a low red blood cell count).

If the patient has a procedure where tumor samples are obtained, like a repeat bone marrow evaluation or tumor biopsy, the investigators request a sample to be used for research purposes. Patients will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
1. INCLUSION CRITERIA AT TIME OF PROCUREMENT

   1. Any patient, regardless of age or sex, with EBV-positive Hodgkin's or non Hodgkin's Lymphoma, (regardless of the histological subtype) or EBV (associated)- T/NK-lymphoproliferative disease who may subsequently be eligible for the treatment component
   2. EBV positive tumor (can be pending)
   3. Weighs at least 10 kg
   4. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given a copy of informed consent.
2. INCLUSION CRITERIA AT TIME OF INFUSION

   1) Any patient regardless of age or sex, with diagnosis of either
   1. EBV positive Hodgkin's lymphoma
   2. EBV positive non-Hodgkin's Lymphoma (regardless of histologic subtype)
   3. EBV (associated)-T/NK-lymphoproliferative disease

   AND either

   A) In first or subsequent relapse or with persistent active disease despite therapy; OR

   B) With active disease if immunosuppressive chemotherapy is contraindicated as determined by the study PI, in consultation with the primary provider as needed, e.g. patients who develop Hodgkin's disease after solid organ transplantation or if the lymphoma is a second malignancy, e.g. a Richter's transformation of CLL.

   2) EBV positive tumor confirmed by pathology

   3) Patients with life expectancy ≥ 6 weeks

   4) Patients with bilirubin ≤ 3x upper limit of normal, AST ≤ 3x upper limit of normal, creatinine ≤ 2x upper limit of normal for age and Hgb ≥ 7.0 (may be a transfused value)

   5) Pulse oximetry of >90% on room air

   6) Patients should have been off other investigational therapy for 4 weeks prior to entry in this study.

   7) Patients with a Karnofsky/Lansky score of ≥ 50

   8) Informed consent explained to, understood and signed by patient/guardian. Patient/guardian given a copy of informed consent.
3. EXCLUSION CRITERIA AT TIME OF PROCUREMENT

   1. Known pregnancy or actively breastfeeding (pregnancy test is not required at the time of procurement).
4. EXCLUSION CRITERIA AT TIME OF INFUSION

   1. Pregnant or breastfeeding
   2. Active and uncontrolled bacterial, viral or fungal infection
   3. Current use of systemic corticosteroids (prednisone equivalent >0.5 mg/kg/day)
   4. Bulky disease resulting in airway obstruction or risk for airway obstruction with further enlargement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2039-03-30 (Estimated)

PRIMARY OUTCOMES:
1. Dose limiting toxicity rate (DLT) by Common Terminology Criteria for Adverse Events v5.0 | 28 days post infusion
  Dose-limiting toxicity is defined as any irreversible, life threatening or non-hematologic Grade 3-5 event considered to be primarily related to the EBVST infusion, with the exception of Grade 3-4 expected reactions such as fever and hypotension/ Grade 3-4 CRS toxicity persistent beyond 72 hours.

SECONDARY OUTCOMES:
1. Response rate by Lymphoma Response to Immunomodulatory Therapy (LYRIC) criteria | 6 weeks (±2 weeks) post infusion
  The response rate is calculated as the percentage of patients whose best response is either complete response or partial response according to Lyric criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Sharma S, Mehta NU, Sauer T, Rollins LA, Dittmer DP, Rooney CM. Cotargeting EBV lytic as well as latent cycle antigens increases T-cell potency against lymphoma. Blood Adv. 2024 Jul 9;8(13):3360-3371. doi: 10.1182/bloodadvances.2023012183. PMID 38640255
- [Derived] Sharma S, Sauer T, Omer BA, Shum T, Rollins LA, Rooney CM. Constitutive Interleukin-7 Cytokine Signaling Enhances the Persistence of Epstein-Barr Virus-Specific T-Cells. Int J Mol Sci. 2023 Oct 31;24(21):15806. doi: 10.3390/ijms242115806. PMID 37958791